CLINICAL TRIAL: NCT05404373
Title: The Efficacy and Safety of Normobaric Hyperoxia on Treatment Duration for Acute Ischemic Stroke Patients With Endovascular Treatment
Brief Title: Treatment Duration on Normobaric Hyperoxia in Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TD-NBO
Record Dates: First submitted 2022-05-24; First posted 2022-06-03 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-06

CONDITIONS: Stroke, Acute; Neuroprotection; Endovascular Treatment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low flow oxygen group (Placebo Comparator): patients were randomized into the Low flow oxygen group and immediately given 100% oxygen inhalation (no more than 30 minutes after admission) at a ventilation rate of 1L/ min using a oxygen storage mask and keep giving oxygen for 4 hours.
  Interventions: Other: Low flow oxygen
- NBO group (2h) (Experimental): patients were randomized into the NBO group (2h) and immediately given 100% oxygen inhalation (no more than 30 minutes after admission) at a ventilation rate of 10L/ min using a oxygen storage mask and keep giving oxygen for 2 hours.
  Interventions: Other: Normobaric Hyperoxia (NBO)
- NBO group (4h) (Experimental): patients were randomized into the NBO group (4h) and immediately given 100% oxygen inhalation (no more than 30 minutes after admission) at a ventilation rate of 10L/ min using a oxygen storage mask and keep giving oxygen for 4 hours.
  Interventions: Other: Normobaric Hyperoxia (NBO)
- NBO group (6h) (Experimental): patients were randomized into the NBO group (6h) and immediately given 100% oxygen inhalation (no more than 30 minutes after admission) at a ventilation rate of 10L/ min using a oxygen storage mask and keep giving oxygen for 6 hours.
  Interventions: Other: Normobaric Hyperoxia (NBO)

INTERVENTIONS:
Other: Normobaric Hyperoxia (NBO) — NBO was inhaled as early as possible before revascularization, and inhaled for 1h/2h/4h according to different groups
  Arms: NBO group (2h); NBO group (4h); NBO group (6h)
Other: Low flow oxygen — immediately given oxygen inhalation at a ventilation rate of 1L/ min using a oxygen storage mask and keep giving oxygen for 4 hours.
  Arms: Low flow oxygen group

SUMMARY:
Normoxia Hyperoxia (NBO) is a neuroprotective approach that can be implemented early. NBO is simple and non-invasive and can be used at home or in an ambulance to ensure the shortest possible time after cerebral ischemia occurs. The previous study by the investigators suggested that NBO therapy in the early stage of cerebral ischemia has a neuroprotective effect on ischemic brain injury. Although the neuroprotective effect of NBO has been demonstrated, the optimal duration of treatment for NBO to exert neuroprotective effect is still unclear. Therefore, further discussion of the duration of NBO treatment will contribute to the clinical application of NBO and provide a definite theoretical basis for the treatment of cerebral infarction.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and signs were consistent with acute anterior circulation stroke,
* NIHSS score≥6分;Alberta Stroke Program Early CT score (ASPECTS)≥6;
* Met the indications for endovascular therapy;
* (Level of consciousness)NIHSS score 0 or 1; MRS score was 0-1 before stroke
* The time from onset to randomization was within 24 hours;
* Preoperative CTA or MRA confirmed the presence of large vessel occlusion (internal carotid artery or middle cerebral artery M1, M2 segments);
* Patients and their families signed informed consent

Exclusion Criteria:

* Rapid neurological function improvement, NIHSS score less than 10 points, or evidence of vessel recanalization prior to randomization;
* Seizures at stroke onset;
* Intracranial hemorrhage;
* Symptoms suggestive of subarachnoid hemorrhage, even if CT scan was normal;
* Known hemorrhagic diathesis, coagulation factor deficiency, or on anticoagulant therapy with INR > 3.0 or PTT > 3 times normal;
* Platelet count of less than 100,000 per cubic millimeter;
* Severe hepatic or renal dysfunction;
* Severe, sustained hypertension (Systolic Blood Pressure >185 mmHg or Diastolic Blood Pressure >110 mmHg)
* Baseline blood glucose of <50mg/dL (2.78 mmol) or >400mg/dL (22.20 mmol) Active and chronic obstructive pulmonary disease or acute respiratory distress syndrome;
* >3 L/min oxygen required to maintain peripheral arterial oxygen saturation (SaO2) 95% as per current stroke management guidelines;
* Medically unstable;
* Life expectancy<90 days;
* Patients who could not complete the 90-day follow-up;
* Evidence of intracranial tumor;
* Patients with anemia or polycythemia vera or other situations that require urgent oxygen inhalation;
* Patients with upper gastrointestinal bleeding or nausea or vomiting so that they cannot cooperate with the mask to inhale oxygen.
* A history of severe allergies to contrast agents;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Cerebral infarct volume | Within 72 hours after randomization
  The infarct volume is evaluated by MRI or CT scan

SECONDARY OUTCOMES:
Scores assessed by National Institutes of Health Stroke Scale(NIHSS) | 24hours, 72hours, day7 after randomization
  secondary clinical efficacy endpoint; the NIHSS is a stroke severity score composed of 11 items (range from 0 to 41, higher values indicate more severe deficits)
The proportion of good prognosis | 90 ± 10 days after randomization
  the mRs is an ordinal disability score of 7 categories (0 = no symptoms to 5 = severe disability, and 6 = death;with higher scores indicating more severe disability);The ratio of 0 to 2;
neurological function improvement rate | Time Frame: 24 ± 6 hours
  NIHSS score increased by more than 4 points);the NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits);
modified Rankin Scale score (mRS) score | 30 ± 7 days, 90 ± 10 days after randomization;
  secondary clinical efficacy endpoint; the mRs is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability,and 6=death)
Vascular recanalization rate | Time Frame: 4 hours ± 15 minutes
  secondary imaging efficacy endpoint; Extended Treatment In Cerebral Ischemia (eTICI)；The eTICI is an ordinal hierarchical scale ranging from 0 to 3, with higher scores indicating better antegrade reperfusion of the previously occluded target artery ischemic territory; eTICI 2B or 3 are defined as successful recanalization;
blood biomarkers : occludin(ng/ml), MMP-9(ng/ml), S100B(ng/ml),NSE(ng/ml),GFAP(ng/ml),PGP9.5(ng/ml),etc | 24 ± 6 hours, 72 ± 24 hours
  Biomarkers for evaluation of BBB damage , brain injury and inflammation,etc:
Incidence of oxygen-related adverse events | 24 ± 6 hours,
  Including Headache, dizziness, nausea, vomiting, chest tightness, shortness of breath, cough,etc;
Incidence of neurologic deterioration; | 24 ± 6 hours;
  NIHSS score increased by more than 4 points);the NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits);clinical safety endpoint;
Incidence of Symptomatic Intracerebral Hemorrhage | 24± 12 hours hours after randomization
  imaging safety endpoints;Deterioration in NIHSS score of ≥4 points within 24 hours;per ECASS III definition and per Heidelberg bleeding classification
Incidence of any intracranial hemorrhage | 24± 12 hours hours after randomization
  imaging safety endpoints;per ECASS III definition and per Heidelberg bleeding classification
all-cause death rate | 90 ± 10 days after randomization
  clinical safety endpoint; Ratio of total deaths from all causes to all enrollments
Incidence of adverse events | 90 ± 10 days after randomization
  clinical safety endpoint;
Incidence of surgery-related complications | 24± 12 hours hours after randomization
  clinical safety endpoint;
stroke related death rate | 90 ± 10 days after randomization;
  clinical safety endpoint; Stroke-related deaths as a proportion of all participants
Vital signs:respiration(times/min) | 0 hours, 2 hours, 4 hours after randomization;
  clinical safety endpoint;
Vital signs:heart rate: (times/min) | 0 hours, 2 hours, 4 hours after randomization;
  clinical safety endpoint;
Vital signs:blood pressure(mmHg) | 0 hours, 2 hours, 4 hours after randomization;
  clinical safety endpoint;
Vital signs:oxygen saturation (%) | 0 hours, 2 hours, 4 hours after randomization;
  clinical safety endpoint;

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Li W, Wang S, Liu L, Chen J, Lan J, Ding J, Chen Z, Yuan S, Qi Z, Wei M, Ji X. Normobaric Hyperoxia Combined With Endovascular Treatment Based on Temporal Gradient: A Dose-Escalation Study. Stroke. 2024 Jun;55(6):1468-1476. doi: 10.1161/STROKEAHA.123.046106. Epub 2024 May 15. PMID 38747162